CLINICAL TRIAL: NCT00221403
Title: Placebo Controlled Trial of Valproate and Risperidone in Young Children With Bipolar Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-0835
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Bipolar Disorder
Keywords: child; adolescent; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Risperidone; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Valproate (VPA) (Active Comparator): VPA was administered in liquid form, matched for taste and color with the placebo. Medication was administered in a double-blinded manner on a twice-daily basis. Patients randomized to VPA were administered an initial dose of 10 mg/kg/day on a twice daily schedule beginning on day 0. VPA levels were adjusted to achieve a blood level of 80-100 lg/mL. An independent, unblinded study psychiatrist adjusted VPA doses to achieve a therapeutic level
  Interventions: Drug: Valproate Oral Solution
- Risperidone (Active Comparator): Risperidone was administered in liquid form matched for taste and color to the placebo. Medications were administered in a double-blinded manner on a twice-daily basis.
  Interventions: Drug: Risperidone oral solution
- Placebo (Placebo Comparator): The placebo was administered in liquid form, matched for taste and color with the active comparator.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Risperidone oral solution — liquid, BID dosing.
  Other Names: Risperdal
  Arms: Risperidone
Drug: Valproate Oral Solution — liquid, BID dosing.
  Other Names: VPA
  Arms: Valproate (VPA)
Other: Placebo — liquid, BID dosing.
  Arms: Placebo

SUMMARY:
The primary aim of this proposal is to conduct a preliminary controlled trial of valproate and risperidone in children ages 3-7 yr. with bipolar disorders. A secondary aim is to carefully characterize these subjects using clinical rating scales and develop pilot data on a very young cohort of children with bipolar disorders that can be used to support an application to NIMH for a prospective, longitudinal study that will provide important information about the course, medication response, neurobiology and outcome of these patients.

DETAILED DESCRIPTION:
It is now recognized that pediatric bipolar disorders are highly prevalent and that they seriously disrupt the lives of children and adolescents, with studies showing poorer academic performance, disturbed interpersonal relationships, increased rates of substance abuse, legal difficulties, multiple hospitalizations, and increased rates of both suicide attempts and completions (Akiskal, Downs et al. 1985; Lewinsohn, Klein et al. 1995; Strober, Schmidt-Lackner et al. 1995). We are seeing an increasing number of very young children, ages 3-7 years, with either frank symptoms of BP I disorder. Over 50% of these young patients have a first-degree relative with a bipolar disorder and all of these patient's families are significantly impacted by their BP symptoms. Many of these young BP patients have been treated with stimulants or antidepressants and few have been treated with mood stabilizing agents. Therefore, it is necessary to provide controlled studies of psychotropics in this younger bipolar population to provide clinical practice with an appropriate evidence-base.

Several major questions exist about these very young bipolar patients:

* What is the response of these very young bipolar patients to mood stabilizers and or atypical antipsychotics?
* Will non-responders to mono-therapy with either valproate or risperidone respond to treatment with both agents?
* How can we best characterize these patients clinically?
* What is the long-term outcome of these patients?
* Will earlier treatment lead to better outcomes?

The clinical use of mood stabilizers and atypical antipsychotic agents in children and adolescents with bipolar disorders has increased significantly over the past few years, despite the fact that only limited research has suggested that these agents are effective in this population. Common clinical practice is to have patients continue on medications for some time following remission, although the length of continuation treatment varies and available guidelines are based on consensus, not controlled trials. The increased number of medications prescribed has led to concern about over prescribing of psychotropics in children and adolescents (Zito, Safer et al. 2000; Zito, Safer et al. 2003). Therefore, it is necessary to provide additional controlled studies of mood stabilizing agents in this younger bipolar population to guide clinical practice.

There is an overwhelming need for controlled trials of the various mood stabilizers and atypical antipsychotics that are now available and being used in the community with these young bipolar patients. Currently, we have the most experience with valproate and risperidone in bipolar children, ages 8 - 17 yr. and based on clinical experience, believe that these two agents are the safest and most likely to be efficacious in children ages 3-7 years. These agents are widely used in the community and controlled data are desperately needed regarding the effectiveness of these agents in bipolar children, ages 3-7 years. There are no specific behavioral treatments or psychotherapies that have been shown to be efficacious for these patients.

Power Analysis (Provided by Dr. Judy Bean)

Since this is a preliminary study prior to a larger controlled trial, the percent of responders receiving one of the drugs will be compared to the percent of responders in the placebo arm. The children will be randomized to achieve 24 total children in each drug arm and 12 in the placebo arm. This 2:2:1 randomization scheme was selected because the expectation is that the percent of responders, in each of the drug arms, will be greater than the percent in the placebo arm. The expectation is that 60% of the children receiving risperidone will respond (Frazier, Meyer et al. 1999), as compared to only 8% in the placebo group (Geller, Cooper et al. 1998). Power was calculated for a one-sided test since if placebo does better no application will be made to NIH. Using nQuery®, version 5.0, a chi-square test, with a 0.05 significance level, will have 96% power to detect the difference. For valproate, the percent of responders is expected to be 55%(Kowatch, Suppes et al. 2000), as compared to the 8% in the placebo arm. Again, using a chi-square test with a .05 significance level, the power will be 86 with 24 in the valproate arm and 12 in the placebo arm. This pilot study does not power to determine if the two drug arms are equivalent.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 3-7 years 11 months of age.
2. Each patient's authorized legal guardian must understand the nature of the study and must provide written informed consent. Each patient must also give assent to study participation.
3. Patients must have a diagnosis of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) bipolar disorder and must currently display an acute manic, hypomanic or mixed episode as determined by DSM-IV criteria. This includes the following diagnoses: 296.4x, Bipolar I Disorder, Most Recent Episode Manic; 296.6x, Bipolar I Disorder, Most recent Episode Mixed; and 296.0x, Bipolar I Disorder, Single Manic Episode, Bipolar II Disorder, Most Recent Episode Hypomanic.
4. Patients must have an initial score (at day 0) on the YMRS total score of at least 20.
5. Subjects and their caretakers should be fluent in English.

Exclusion Criteria:

1. Clinically significant or unstable hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, hematologic or other systemic medical conditions.
2. Neurologic disorders including epilepsy, stroke, or severe head trauma.
3. Clinically significant laboratory abnormalities, on any of the following tests: CBC with differential, electrolytes, BUN, creatinine, hepatic transaminases, urinalysis, thyroid indices (T3, Total T4, Free T4, TSH), and EKG.
4. Mania due to a general medical condition or substance-induced mania (DSM-IV).
5. Mental retardation (IQ <70), evidence of Fetal Alcohol Syndrome or an Alcohol-Related Neurodevelopmental Disorder.
6. History of hypersensitivity to or intolerance of risperidone or valproate.
7. Prior history of risperidone or valproate non-response.
8. Judged clinically to be at serious suicidal risk.
9. Participation in a clinical trial of another investigational drug within 1 month (30 days) prior to study entry.
10. Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections and day 0.

    -

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2004-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Kowatch, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Kowatch RA, Scheffer RE, Monroe E, Delgado S, Altaye M, Lagory D. Placebo-controlled trial of valproic Acid versus risperidone in children 3-7 years of age with bipolar I disorder. J Child Adolesc Psychopharmacol. 2015 May;25(4):306-13. doi: 10.1089/cap.2014.0166. PMID 25978742

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone: Subjects only taking Risperidone.
- Valproate: Subjects taking Valproate only.
- Placebo: Subjects taking Placebo only.
Period: Overall Study
Arm/Group | Risperidone | Valproate | Placebo
Started | 18 | 21 | 7
Completed | 16 | 16 | 7
Not Completed | 2 | 5 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Risperidone: Subjects taking Risperidone only.
- Total: Total of all reporting groups
Arm/Group | Risperidone | Valproate | Placebo | Total
Number analyzed (Participants) | 18 | 21 | 7 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 21 | 7 | 46
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.31 (1.3) | 6.03 (1.3) | 5.19 (1.0) | 5.51 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 2 | 17
  Male | 11 | 13 | 5 | 29
Region of Enrollment [Number; unit: participants]
  United States | 18 | 21 | 7 | 46

OUTCOME MEASURES:

1. Primary Outcome: YMRS
Description: Young Mania Rating Scale (YMRS) total scores change from baseline by treatment group. The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms.
Time Frame: 6 weeks
Population: Subjects were male or female outpatient subjects, 3.0-7 years,11 months of age, with bipolar I disorder, mixed or manic episode, psychotic or nonpsychotic, according to DSM IV-TR criteria, with a score ‡ 20 (considered to be moderate severity) on the Young Mania Rating Scale (YMRS) at the time of randomization.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valproate (VPA) | Risperidone | Placebo
Number analyzed (Participants) | 21 | 18 | 7
score on a scale | 10 (2.46) | 18.82 (1.55) | 4.29 (3.56)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: AEs were assessed with a checklist (SEFCA), rated on a scale of ''not present'' to ''mild, does not interfere with functioning,'' ''moderate, some interference with functioning,'' and ''severe, functioning is significantly impaired because of side effects.'' A significant AE was identified if not been present at baseline, but was reported during the course of the study, or if it had been present at baseline, but its severity was increased by at least 1 point on the scale during the study.
Arm/Group | Risperidone | Valproate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/21 | 0/7
Other Adverse Events (participants affected / at risk) | 0/18 | 1/21 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone (N=18) | Valproate (N=21) | Placebo (N=7)
nausea (General disorders) | 0 (0) | 1 (1) | 0 (0) — upset stomach

LIMITATIONS AND CAVEATS:
This study was limited by the small sample size and short duration of treatment. The average VPA level of 81 lg/ml was relatively low, and may have limited the response rate to VPA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No